CLINICAL TRIAL: NCT01181726
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fed, Bioequivalence Study of Estradiol/Norethindrone Acetate Tablets, 1 mg/0.5 mg Versus Activella® (1 mg Estradiol/0.5 mg Norethindrone Acetate) Tablets in Normal, Healthy, Post-Menopausal Female Subjects.
Brief Title: Estradiol/Norethindrone Acetate Tablets, 1/0.5 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3252
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — estradiol, norethindrone drug combination; Estradiol; Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): Estradiol/Norethindrone Acetate Tablets, 1 mg/0.5 mg
  Interventions: Drug: Estradiol/Norethindrone acetate
- Reference Listed Drug (Active Comparator): Activella® (1 mg estradiol/0.5 mg norethindrone acetate) Tablets
  Interventions: Drug: Activella®

INTERVENTIONS:
Drug: Estradiol/Norethindrone acetate — 1 mg/0.5 mg Tablets
  Other Names: Mimvey®
  Arms: Investigational Test Product
Drug: Activella® — 1 mg/0.5 mg Tablets
  Other Names: Estradiol/Norethindrone acetate (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The objective of this study was to determine and compare the rate and extent of absorption of norethindrone and unconjugated estradiol from a test formulation of Estradiol/Norethindrone Acetate Tablets, 1 mg/0.5 mg versus the reference Activella® (1 mg estradiol/0.5 mg norethindrone acetate) Tablets under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking (up to 10 cigarettes/day), physiologically or surgically post-menopausal female within the age range of 18-65 years.
* 17β-estradiol serum levels of ≤ 92 pmol/L and follicle-stimulating hormone (FSH) of ≥ 40 IU/L.
* Body Mass Index (BMI) greater than or equal to 19.0 kg/m2 and less than or equal to 30.0 kg/m2.
* Normal findings in the physical examination, 12-lead electrocardiogram (ECG) and vital signs.
* Hemoglobin ≥ 115 g/L.
* Normal pap smear.
* Normal mammogram within 1 year for subjects who are over the age of 50 years.
* Negative for drugs of abuse and alcohol.
* Negative for hepatitis B-surface antigen, hepatitis C, and Human Immunodeficiency Virus (HIV).
* No clinical laboratory values outside the acceptable range unless the Principal Investigator or Sub-Investigator decides that they are not clinically significant (NCS).
* Negative for pregnancy.
* Subjects who are surgically post-menopausal with an intact uterus (i.e. bilateral oophorectomy) for at least 6 months, or physiologically post-menopausal (i.e. spontaneous amenorrhea) for at least 1 year, and who will adhere to contraceptive requirements from at least 10 days before Period I check-in, during the study and up until 1 month after the end of the study.
* Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed ICF.

Exclusion Criteria:

* Known history of hypersensitivity to norethindrone and estradiol combinations and/or norethindrone, and/or estradiol.
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, or hematological diseases, malignancies, or migraines, unless deemed not clinically significant by the Principal Investigator or Sub-Investigator.
* Known history of liver, kidney, and/or gallbladder dysfunction/disease, chronic diarrhea, or inflammatory bowel diseases.
* Known history or presence of cerebrovascular diseases or venous thromboembolic events, including deep vein thrombosis, pulmonary embolism, and retinal vein thrombosis.
* Any history of stroke.
* Presence of any significant physical or organ abnormality.
* History of osteoporosis.
* History or presence of fibrocystic breast disease.
* History or presence of breast, endometrial, cervical, and/or uterine carcinoma.
* Any illness during the 4 weeks before this study, unless deemed not clinically significant by the Principal Investigator or Sub-Investigator.
* Any history or evidence of psychiatric or psychological disease, unless deemed not clinically significant by the Principal Investigator or the Sub-Investigator.
* Any history or abnormal vaginal bleeding, unless deemed not clinically significant by the Principal Investigator or the Sub-Investigator.
* Any history of asthma (after 12 years of age).
* Evidence of pregnancy or lactation.
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Any history or drug abuse.
* Any recent history of alcohol abuse (less than 1 year).
* Use of any prescription medication within 30 days preceding this study.
* Use of hormone replacement therapy within 30 days before drug administration.
* Use of over-the-counter (OTC) medication or any herbal supplement within the 7 days preceding this study.
* Use of hormonal contraceptives, oral, transdermal, implant within 30 days before drug administration or a depot injection or progestogen drug within 1 year before the drug administration.
* Depot injection of any drug within 6 months.
* Blood draws within 56 days preceding this study, during the conduct of any clinical study at another facility, or within the lockout period specified by previous study.
* Blood donations within 56 days preceding this study.
* Participation as a plasma donor in a plasmapheresis program within 7 days preceding this study.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Intolerance to venipuncture.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Tam, M.D., F.R.C.P., F.A.C.P., Principal Investigator — Biovail Clinical Research
Locations (1):
- Biovail Contract Research, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol/Norethindrone Acetate (Test) First: 1 mg/0.5 mg Estradiol/Norethindrone Acetate Tablets test product dosed in first period followed by 1 mg/0.5 mg Activella® Tablets reference product dosed in the second period.
- Activella® (Reference) First: 1 mg/0.5 mg Activella® Tablets reference product dosed in first period followed by 1 mg/0.5 mg Estradiol/Norethindrone Acetate Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Estradiol/Norethindrone Acetate (Test) First | Activella® (Reference) First
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout of 28 Days
Arm/Group | Estradiol/Norethindrone Acetate (Test) First | Activella® (Reference) First
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Estradiol/Norethindrone Acetate (Test) First | Activella® (Reference) First
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol/Norethindrone Acetate (Test) First | Activella® (Reference) First | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 15 | 28
  Hispanic | 3 | 1 | 4
  Black | 2 | 2 | 4
  Asian | 2 | 1 | 3
  American Indian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Norethindrone (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Norethindrone Cmax.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Estradiol/Norethindrone Acetate (Test): 1 mg/0.5 mg Estradiol/Norethindrone Acetate Tablets test product dosed in either period.
- Activella® (Reference): 1 mg/0.5 mg Activella® Tablets reference product dosed in either period.
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
ng/mL | 6.54 (3.62) | 6.06 (2.95)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 104.66, 90% CI 2-sided [94.22 to 116.25] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Norethindrone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Norethindrone AUC0-t.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
ng*h/mL | 45.03 (21.76) | 46.13 (21.62)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.4, 90% CI 2-sided [93.91 to 101.02] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Norethindrone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Norethindrone AUC0-inf.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
ng*h/mL | 49.55 (23.08) | 50.68 (22.78)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.60, 90% CI 2-sided [94.05 to 101.30] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Corrected Total Estrone(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Corrected Total Estrone Cmax.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 27076.08 (11600.13) | 27240.03 (11610.70)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.35, 90% CI 2-sided [92.21 to 107.06] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: AUC0-t of Corrected Total Estrone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on Corrected Total Estrone AUC0-t.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 384547.68 (185543.06) | 407028.98 (191192.18)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 95.21, 90% CI 2-sided [91.21 to 99.39] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: AUC0-inf of Corrected Total Estrone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on Corrected Total Estrone AUC0-inf.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 380131.12 (163543.17) | 424801.99 (216597.41)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 95.25, 90% CI 2-sided [91.18 to 99.51] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Cmax of Uncorrected Total Estrone(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for Uncorrected Total Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 27256.41 (11652.78) | 27430.77 (11674.97)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.33, 90% CI 2-sided [92.21 to 107.00] — This analysis was for informational purposes only and was not used to establish bioequivalence

8. Secondary Outcome: AUC0-t of Uncorrected Total Estrone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for Uncorrected Total Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 397537.88 (193337.67) | 420763.02 (198975.61)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 95.19, 90% CI 2-sided [91.18 to 99.38] — This analysis was for informational purposes only and was not used to establish bioequivalence

9. Secondary Outcome: AUC0-inf of Uncorrected Total Estrone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for Uncorrected Total Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 398139.63 (173723.79) | 425739.45 (198546.75)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 95.23, 90% CI 2-sided [91.17 to 99.47] — This analysis was for informational purposes only and was not used to establish bioequivalence

10. Secondary Outcome: Cmax of Uncorrected Unconjugated Estradiol(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for Uncorrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 59.24 (19.10) | 60.33 (19.04)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.92, 90% CI 2-sided [93.44 to 102.61] — This analysis was for informational purposes only and was not used to establish bioequivalence

11. Secondary Outcome: AUC0-t of Uncorrected Unconjugated Estradiol(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for Uncorrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 2016.26 (596.40) | 2086.39 (746.24)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.77, 90% CI 2-sided [93.92 to 101.78] — This analysis was for informational purposes only and was not used to establish bioequivalence

12. Secondary Outcome: AUC0-inf of Uncorrected Unconjugated Estradiol(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for Uncorrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 2301.59 (642.09) | 2274.04 (784.48)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.71, 90% CI 2-sided [94.42 to 105.30] — This analysis was for informational purposes only and was not used to establish bioequivalence

13. Secondary Outcome: Cmax of Uncorrected Unconjugated Estrone(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for Uncorrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 513.56 (165.85) | 529.23 (217.12)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.19, 90% CI 2-sided [94.71 to 103.87] — This analysis was for informational purposes only and was not used to establish bioequivalence

14. Secondary Outcome: AUC0-t of Uncorrected Unconjugated Estrone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for Uncorrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 12444.22 (4018.39) | 12977.00 (5291.36)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.83, 90% CI 2-sided [94.55 to 101.21] — This analysis was for informational purposes only and was not used to establish bioequivalence

15. Secondary Outcome: AUC0-inf of Uncorrected Unconjugated Estrone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for Uncorrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 13592.44 (3686.14) | 14155.46 (5300.06)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 98.01, 90% CI 2-sided [94.54 to 101.60] — This analysis was for informational purposes only and was not used to establish bioequivalence

16. Secondary Outcome: Cmax of Corrected Unconjugated Estradiol(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for Corrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 55.18 (19.31) | 56.24 (19.26)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.87, 90% CI 2-sided [93.22 to 102.74] — This analysis was for informational purposes only and was not used to establish bioequivalence

17. Secondary Outcome: AUC0-t of Corrected Unconjugated Estradiol(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for Corrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 1723.44 (540.76) | 1793.04 (689.12)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.96, 90% CI 2-sided [93.66 to 102.46] — This analysis was for informational purposes only and was not used to establish bioequivalence

18. Secondary Outcome: AUC0-inf of Corrected Unconjugated Estradiol(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for Corrected Unconjugated Estradiol.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 1823.43 (551.11) | 1871.56 (730.51)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.01, 90% CI 2-sided [94.17 to 104.11] — This analysis was for informational purposes only and was not used to establish bioequivalence

19. Secondary Outcome: Cmax of Corrected Unconjugated Estrone(Maximum Observed Concentration of Drug Substance in Plasma)
Description: Informational comparison of Cmax values for Corrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg/mL | 492.81 (166.57) | 509.81 (217.80)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.13, 90% CI 2-sided [94.39 to 104.10] — This analysis was for informational purposes only and was not used to establish bioequivalence

20. Secondary Outcome: AUC0-t of Corrected Unconjugated Estrone(Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Informational comparison of AUC0-t values for Corrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 10952.25 (3887.84) | 11369.60 (5058.92)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.72, 90% CI 2-sided [94.03 to 101.56] — This analysis was for informational purposes only and was not used to establish bioequivalence

21. Secondary Outcome: AUC0-inf of Corrected Unconjugated Estrone(Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Informational comparison of AUC0-inf values for Corrected Unconjugated Estrone.
Time Frame: Blood samples collected over a 72 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Number analyzed (Participants) | 39 | 39
pg*h/mL | 11293.21 (3899.12) | 11747.97 (5289.05)
Statistical Analysis 1: Comparison: Estradiol/Norethindrone Acetate (Test) vs Activella® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 97.99, 90% CI 2-sided [94.11 to 102.02] — This analysis was for informational purposes only and was not used to establish bioequivalence

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Estradiol/Norethindrone Acetate (Test) | Activella® (Reference)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol/Norethindrone Acetate (Test) (N=40) | Activella® (Reference) (N=40)
Headache (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.